CLINICAL TRIAL: NCT06742632
Title: Comparative Study in Psychiatric Problems Among Mothers With Miscarriage in First and Second Trimester
Brief Title: Comparative Psychiatric Problems Between First and Second Trimester Miscarriage
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer of psychiatry,assiut university, Assiut University
Other Study IDs: psychiatry issues in Abortion
Record Dates: First submitted 2024-12-11; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Abortion
Keywords: abortion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- first trimester abortion
  Interventions: Behavioral: Symptoms checklist-90
- second trimester abortion
  Interventions: Behavioral: Symptoms checklist-90

INTERVENTIONS:
Behavioral: Symptoms checklist-90 — The Symptom Checklist-90 (SCL90) is a 90-item questionnaire used to assess psychological problems. The Symptom Checklist-90-Revised (SCL90R) is the revised version of the questionnaire.

SUMMARY:
Description of the psychiatric impact of miscarriage on women.

DETAILED DESCRIPTION:
miscarriage, a significant reproductive health issue, often has profound psychological implications for women. The emotional and psychiatric effects of abortion can vary widely based on individual, cultural, and situational factors, as well as the timing of the procedure (1). First-trimester abortions are typically more common and are generally less complex medically, while second-trimester abortions often involve more intricate decision-making processes and greater societal and personal stigma (2).

Emerging evidence suggests that women undergoing abortions in different trimesters may experience distinct psychiatric challenges, including anxiety, depression, and post-traumatic stress disorder. However, the comparative psychological burden between first- and second-trimester abortions remains underexplored (3-6). Understanding these differences is crucial for tailoring mental health interventions and providing comprehensive care to affected women.

This study aims to compare the prevalence and types of psychiatric problems in mothers undergoing abortion in the first versus the second trimester, thereby contributing to the body of knowledge on maternal mental health and informing evidence-based support strategies.

ELIGIBILITY:
Inclusion Criteria:

* all miscarrying women less than or equal to 26 weeks gestation

Exclusion Criteria:

* ectopic pregnancy and vesicular mole

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: all miscarrying women aged from 28 to 45 years less than or equal to 26 weeks gestation
Sampling Method: Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
measure psychiatric problems among the stuided groups | through study completion, an average of 3 months
  symptom checklist 90 "SCL 90'': It is a 90-item ques tionnaire used to assess psychological problems. Each item is scored on a scale from 0 to 4 based on how much an individual was bothered by each item. It has 9 subscales: (Somatization, Obsessive-compulsive, Inter personal sensibility, Depression, Anxiety, Anger-hostility, Phobic-anxi ety, Paranoid ideation, Psychoticism).

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ayaulym N. Blushinova, Gulnara M. Shalgumbayeva, Duman Berikuly, Zaituna G. Khamidullina, Gaukhar A. Korganbayeva, Inabat N. Ordabayeva, Nazerke K. Sailauova ABB. Epidemiological aspects of pregnant losses. literature review. Sci Healthc J. 2023;25(2):236-43.
- [Result] Herbert D, Young K, Pietrusinska M, MacBeth A. The mental health impact of perinatal loss: A systematic review and meta-analysis. J Affect Disord. 2022 Jan 15;297:118-129. doi: 10.1016/j.jad.2021.10.026. Epub 2021 Oct 20. PMID 34678403